CLINICAL TRIAL: NCT01442116
Title: Evaluation of Regional Myocardial Dynamics at Physical Stress in Essential Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mustafa Kemal University (Other)
Responsible Party: Principal Investigator, Nagehan Kucukler, Principle Investigator, Mustafa Kemal University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: HT60
Record Dates: First submitted 2011-09-15; First posted 2011-09-28 (Estimated); Last update posted 2011-09-29 (Estimated); Status verified 2011-09

CONDITIONS: Hypertension; Left Ventricular Hypertrophy
MeSH Terms: conditions — Hypertension; Hypertrophy, Left Ventricular

ARMS (1):
- Hypertensives (Experimental)
  Interventions: Procedure: stress echocardiography

INTERVENTIONS:
Procedure: stress echocardiography — safety and efficacy of stress echocardiography

SUMMARY:
The study hypothesis is stress-related regional tissue dynamics is related to left ventricular outflow tract blood flow.

ELIGIBILITY:
Inclusion Criteria:

* Essential hypertension

Exclusion Criteria:

* History of Myocardial Infarction
* Diabetes Mellitus
* Renal Failure
* Orthopedic problems

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-06; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
measurement of LVOT velocity before and after exercise by echocardiography | 1 day (before and after exercise stress)
measurement of TDI S wave before and after exercise by echocardiography | 1 day (before and after exercise)

SECONDARY OUTCOMES:
myocardial regional functions measured by tissue Doppler imagination | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Fatih Yalcin, MD, Study Director — Mustafa Kemal University: Turkey
Locations (1):
- Mustafa Kemal University School of Medicine, Department of Cardiology, Antioch, Antioch, Turkey (Türkiye)